CLINICAL TRIAL: NCT02870374
Title: For a Better Interpretation of Quality of Life Scores of Kidney Transplant Patients: Determination of the Minimum Significant Change RetransQol
Acronym: ReTransQol
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-15; 2012-A00634-39 (Other: Ansm)
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Kidneys Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Answering specific quality of life questionnaire in kidneys transplantation population

SUMMARY:
The project team developped and validated a French patient-based health-related quality of life instrument in kidney transplant: the QoL Retrans.

The aim of the study is to determine the minimum significant change of the valdiated tool: ReTransQol

ELIGIBILITY:
Inclusion Criteria:

* Patient with a transplant kidney

Exclusion Criteria:

* Patient not able to answer survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidneys transplanted patients
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-03 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Number of change in quality of life in kidneys transplantation patients using ReTransQol | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille; Stéphanie GENTILE, MD/PhD, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No